CLINICAL TRIAL: NCT01344343
Title: HIP Fracture Accelerated Surgical TreaTment And Care tracK (HIP ATTACK) Trial - Feasibility Pilot
Brief Title: HIP Fracture Accelerated Surgical TreaTment And Care tracK (HIP ATTACK) Trial
Acronym: HIPATTACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, P.J. Devereaux, MD, PhD, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HIPATTACK -6.0, 2012-09-24
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accelerated hip fracture surgery (Experimental): Arrival in the operating room within 6 hours of diagnosis of a hip fracture requiring surgical repair
  Interventions: Other: Accelerated surgical hip fracture repair
- Standard care (No Intervention): Surgical hip fracture repair according to the standard timing

INTERVENTIONS:
Other: Accelerated surgical hip fracture repair — Accelerated hip fracture surgery defined as arrival in the operation room within 6 hours of diagnosis of a hip fracture requiring surgery
  Arms: Accelerated hip fracture surgery

SUMMARY:
There is preliminary evidence that suggests early surgical treatment of a hip fracture may improve patients' outcomes. The investigators propose to do a pilot randomized controlled trial (RCT) to assess the feasibility of a large RCT comparing accelerated surgical repair (i.e. surgery within 6 hours of a hip fracture diagnosis) versus standard care (typically surgery after 36-48 hours).

DETAILED DESCRIPTION:
Hip fractures have devastating consequences: the 30-day mortality rate for men is 9% and for women is 5%, and the risk of disability is substantial. Even among patients who are community-dwelling prior to their hip fracture, 11% are bed-ridden and 16% are in a long-term care facility after one year.

The trauma associated with a hip fracture results in pain, bleeding, and immobility. These factors initiate inflammatory, hypercoaguable, stress, and catabolic states that can cause medical complications, including death. Proposed mechanisms for increased mortality and morbidity associated with delayed surgery include 1) complications related to a protracted immobilization (e.g. venous thromboembolism, atelectasis and pneumonia, urinary tract infections, pressure ulcers, and muscle mass loss) and 2) increased cardiovascular events.

Delay in surgery may result in protracted immobility and the associated complications, as well as prolonged exposure to the hypercoagulable-inflammatory-sympathetic state which may increase cardiovascular events. Observational data suggests that these mechanisms are indeed important: delayed surgical repair is associated with increased mortality and morbidity after a hip fracture.

A systematic review and meta-analysis of observational studies addressed the impact of timing of surgery on the outcome after hip fracture. Five studies reported adjusted measures for mortality. The pooled estimate, based on 721 deaths in 4,208 patients, suggested that early surgical treatment (i.e. within the cut-off of the individual studies) of hip fractures was associated with a significant reduction in mortality (adjusted risk ratio [RR] 0.81, 95% confidence interval [CI] 0.68-0.96).

It is possible that these observational data substantially underestimates the real potential of early surgery. The reason is that the "early surgery" in these studies occurred within 24, 48 or 72 hours. If surgery could be uniformly undertaken within 6 hours, given the potential benefits of earlier mobilization and minimization of the period of the inflammatory hypercoagulable state, the benefits might be substantially greater. The substantial impact of treatment of acute myocardial infarction (MI) or stroke within hours adds credence to this possibility.

Despite the evidence, and the possibility that a larger effect might result from even earlier surgery, current data supports only weak inferences. The evidence relies on observational data and is therefore susceptible to residual confounding. The strength of inference from current evidence does not lay a sufficient solid base to justify the substantial system modification required to facilitate accelerated surgical access for all hip fracture patients.

The main factors that cause surgical delay after a hip fracture are: 1) the patient presents with comorbidities and surgery is deferred for preoperative diagnostics, risk stratification, and medical optimization ("medical clearance") and 2) surgical operating room and staff resources are not available because hip fractures have low priority in urgent surgery lists ("queuing"). Both medical clearance and queuing are modifiable issues - addressing these obstacles has the potential to substantially reduce surgical wait times.

Our ultimate goal is to undertake a large multicentre randomized controlled trial (RCT) of accelerated surgical care (i.e., goal of surgery within 6 hours of diagnosis) versus usual timing of surgery among elderly adults diagnosed with a hip fracture. This protocol is for a pilot RCT that will inform the feasibility of undertaking a large RCT.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 45 years AND
2. diagnosed during working hours on week days with a hip fracture requiring surgery

Exclusion criteria:

We will exclude patients based on the following criteria:

1. patients requiring urgent surgery or urgent interventions for another reason (e.g., subdural hematoma, abdominal pathology requiring urgent laparotomy, acute limb ischemia, other fractures or trauma requiring urgent surgery, or necrotising fascitis; PCI; pacemaker-implantation);
2. open hip fracture;
3. patients refusing participation;
4. patients previously enrolled in the study;
5. Therapeutic anticoagulation not induced by warfarin or intravenous heparin.

Criteria in which the timeline of the surgery in the accelerated care group (after accelerated medical work-up) are at the discretion of the attending physicians.

1. acute myocardial infarction associated with a mechanical complication (i.e., acute papillary muscle rupture, ventricular septal defect) or ST-elevation MI;
2. cardiac arrest;
3. cardiogenic shock, defined by systemic hypotension and symptoms of organ hypoperfusion (oliguria, change in mental status, cold extremities) that the treating physician believes is due to a low cardiac output state (measurement of cardiac index or pulmonary capillary wedge pressure is not required) or requiring inotropic drugs;
4. frank pulmonary edema that cannot be corrected within 2 hours (i.e. after 2 hours the patient cannot maintain oxygen saturation ≥ 90% in supine position with nasal oxygen or 28% oxygen);
5. respiratory failure requiring mechanical ventilation;
6. known pulmonary artery hypertension (> 80 mm Hg);
7. home oxygen therapy with concomitant non-warfarin full dose anticoagulation or clopidogrel (because regional anesthesia is not possible);
8. presumptive bacteremia on the basis of fever ≥ 39° Celsius or two of the following: a) Temperature >38° Celsius or <35° Celsius; b) WBC >12 or < 4 or >10% immature bands; c) rigors; and d) hypotension with evidence of organ dysfunction;
9. hereditary or acquired coagulopathy that cannot be corrected within 2 hours to a INR < 1.5,
10. thrombocytopenia (platelets < 75) of unknown origin that cannot be corrected within 2 hours or in case of known chronic thrombocytopenia platelets < 50;
11. deep venous thrombosis in the last month requiring implantation of vena-cava filter;
12. acute stroke within 7 days of fracture;
13. subarachnoid hemorrhage within 1 month of fracture;
14. impaired consciousness of unknown origin (Glasgow coma scale < 12);
15. fractures acquired during a seizure in patients without a known history of epilepsy;
16. hyponatremia (< 120 mmol/L) or hypernatremia (> 155 mmol/L) or hyponatremia < 125 mmol/L or hypernatremia >150 mmol/L associated with severe neurological symptoms (impaired consciousness to coma, seizures);
17. hyperkalemia > 5.5 mmol/L with QRS-complex > 120 milliseconds (in patients without known previous QRS-complex > 120 ms) or hypokalemia < 2.8 mmol/L not amenable to correction within 2 hours;
18. known pH < 7.15 not amenable to correction within 2 hours; or
19. indication for acute dialysis.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Feasibility | 18 months
  Feasibility defined as:
  * ability to recruit 60 patients in 18 months
  * ability to achieve arrival in the operating room within 6 hours of diagnosis in >=80% of the patients randomized to accelerated surgery
  * ability to achieve accelerated surgery in a timely manner
  * ability to achieve medical clearance in a timely manner
  * resource requirements to achieve recruitment and follow up

SECONDARY OUTCOMES:
All-cause mortality | 30 days
Length of hospital stay | 30 days
Length of intensive care unit stay | 30 days
Length of stay in rehabilitation facility | 30 days
New admission to a long-term care facility | 30 days
Functional Independence Measure (motor domain) | 30 days
Short form health survey (SF-36) (acute form) | 30 days
  Acute form = 1 week recall
Delirium | 7 days after randomization
  Delirium, as defined by the Confusion Assessment Method
Pre-operative Myocardial Infarction | 30 Days
Nonfatal Stroke | 30 Days
Nonfatal Pneumonia | 30 Days
Nonfatal Pulmonary Embolism | 30 Days
Sepsis | 30 Days
New Congestive Heart Failure | 30 Days
Nonfatal Cardiac Arrest | 30 Days
Nonfatal myocardial injury after non cardiac surgery (MINS) | 30 Days
  Myocardial cell injury caused by ischemia, which occurs within 30 days after noncardiac surgery and has short-term prognostic relevance.
  The diagnostic criteria for MINS is within the first 30-days after noncardiac surgery a troponin T value ≥0.03 ng/mL that is felt do to ischemia. MINS does not include perioperative myocardial injury that is due to pulmonary embolism, sepsis, cardioversion, a known troponin antibody or known chronically elevated troponin measurements, or another known nonischemic etiology.
Composite Endpoint | 30 Days
  Composite Outcome of of all-cause mortality, nonfatal pre-operative myocardial infarction, nonfatal myocardial injury after noncardiac surgery (MINS), nonfatal pulmonary embolism, nonfatal pneumonia, nonfatal life-threatening or major bleeding, and nonfatal stroke at 30 days.
Major or Life-threatening Bleeding | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Devereaux, MD, PhD, Principal Investigator — Population Health Research Institute, McMaster University; Mohit Bhandari, MD, MSc, Principal Investigator — Hamilton Health Sciences Corporation
Locations (3):
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph Healthcare Hamilton, Hamilton, Ontario
- Sancheti Institute for Orthopaedics and Rehabilitation, Pune, Maharashtra, India

REFERENCES:
- [Background] Simunovic N, Devereaux PJ, Sprague S, Guyatt GH, Schemitsch E, Debeer J, Bhandari M. Effect of early surgery after hip fracture on mortality and complications: systematic review and meta-analysis. CMAJ. 2010 Oct 19;182(15):1609-16. doi: 10.1503/cmaj.092220. Epub 2010 Sep 13. PMID 20837683
- [Derived] Hip Fracture Accelerated Surgical Treatment and Care Track (HIP ATTACK) Investigators. Accelerated care versus standard care among patients with hip fracture: the HIP ATTACK pilot trial. CMAJ. 2014 Jan 7;186(1):E52-60. doi: 10.1503/cmaj.130901. Epub 2013 Nov 18. PMID 24246589